CLINICAL TRIAL: NCT00880321
Title: A Phase I, Open-Label, Multiple-Dose, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of the BRAF Inhibitor GSK2118436 in Subjects With Solid Tumors
Brief Title: A Phase I Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of GSK2118436 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112680
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: first time in human; BRAF inhibitor; dose escalation
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Part 1 will identify the recommended Part 2 dose using a dose-escalation procedure. Escalation may proceed until either a maximum tolerated dose is established, or the toxicokinetic safety limit is reached. Subjects may dose up to three times a day.
  Interventions: Drug: GSK2118436
- Part 2 (Experimental): Part 2 will explore further the safety, tolerability, and clinical activity of GSK2118436 in subjects with BRAF mutation-positive tumors using the recommended part 2 dose identified during Part 1. Biologically active doses will be identified by measurement of pharmacodynamic markers in tumor tissue and blood across a range of doses and these doses may be explored in Part 2.
  Interventions: Drug: GSK2118436; Drug: Midazolam

INTERVENTIONS:
Drug: GSK2118436 — Dose escalation with GSK2118436 may proceed until either a maximum tolerated dose is established, or the toxicokinetic safety limit is reached.
  Arms: Part 1
Drug: GSK2118436 — Part 2 will use the recommended Part 2 dose of GSK2118436 identified during Part 1 of the study. Biologically active doses will be identified by measurement of pharmacodynamic markers in tumor tissue and blood across a range of doses and these doses may be explored in Part 2.
  Arms: Part 2
Drug: Midazolam — Midazolam will be administered alone and with GSK2118436 in a sub-set of subjects in Part 2 to study the effect of GSK2118436 on CYP3A using midazolam as a probe.
  Arms: Part 2

SUMMARY:
BRF112680 is a first-time-in-human study to establish the recommended dose and schedule of the orally administered GSK2118436. The recommended dose and regimen will be selected based on the safety, pharmacokinetic, and pharmacodynamic profiles observed after the treatment of subjects with solid tumors. This is a two-part study. Part 1 will identify the recommended Part 2 dose using a dose-escalation procedure. Escalation may proceed until either a maximum tolerated dose is established, or the toxicokinetic safety limit is reached. The recommended Part 2 dose will be expanded to up to 12 patients. Part 2 will explore further the safety, tolerability, and clinical activity of GSK2118436 in subjects with BRAF mutation-positive tumors. In addition, the effect of GSK2118436 on midazolam will be assessed in a subset of patients in Part 2. Biologically active doses will be identified by measurement of pharmacodynamic markers in tumor tissue and blood across a range of doses and these doses may be explored in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* 18 years old or older. Subjects enrolled in the midazolam cohort need to be younger than 65 years old.
* Histologically or cytologically confirmed diagnosis of a solid tumor that is not responsive to standard therapies or for which there is no approved or curative therapy. Subjects must have BRAF mutant positive tumors.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain oral medication.
* Male subjects must agree to use one of the contraception methods listed in the protocol. The criterion must be followed from the time of the first dose of study medication until 16 weeks after the last dose of study medication.
* A female subject is eligible to participate if she is of non-childbearing potential or postmenopausal as defined in the protocol. A female of child-bearing potential may participate if she agrees to use one of the contraception methods listed in the protocol.
* Adequate organ system function as defined in the protocol.
* Part 2/Cohorts A, B and C: Must have radiologically and/or clinically documented disease with at least one measurable lesion as defined by RECIST criteria.
* Part 2/Cohort C only: Must have BRAF positive melanoma with the V600E mutation.

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immuno-therapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization).
* Use of an investigational anti-cancer drug within 28 days preceding the first dose of GSK2118436.
* Current use of a prohibited medication as defined in the protocol or requires any of these medications during treatment with GSK2118436.
* Current use of therapeutic warfarin.
* Any major surgery, radiotherapy, or immunotherapy within 4 weeks prior to first dose. Limited radiotherapy within 2 weeks prior to first dose.
* Chemotherapy regimens with delayed toxicity within four weeks prior to first dose (6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within 2 weeks prior to first dose.
* Unresolved toxicity greater than National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0 Grade 1 from previous anti-cancer therapy except alopecia unless agreed to by a GSK Medical Monitor and the investigator.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* A history of known HIV infection.
* Primary malignancy of the central nervous system.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Subjects previously treated for these conditions that are asymptomatic and off corticosteroids for at least two weeks are permitted. Brain metastases must be stable for at least 3 months with verification by imaging (brain MRI completed at screening). Subjects are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs). In Part 2 of the study, subjects with asymptomatic, untreated brain metastases that have not been stable for 3 months may be enrolled with approval of the GSK medical monitor. These subjects can be on a stable dose of corticosteroids.
* History of alcohol or drug abuse within 6 months prior to the screen visit.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
* QTc interval greater than or equal to 480 msecs.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within 24 weeks prior to the first dose.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Abnormal cardiac valve morphology (subjects with minimally abnormalities can be entered on study with approval from the GSK medical monitor).
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, or excipients as described in the protocol (to date there are no known FDA approved drugs chemically related to GSK2118436).
* Pregnant or lactating female.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency.
* Patients positive for HPV. Entry on study allowed only at the discretion of subject and investigator after informed consent regarding discussion of the risk of papillomavirus infection. If enrolled, these subjects must use condoms for sexual activity, regardless of the use of other contraceptive measures and childbearing status.
* Prior treatment with a BRAF or MEK inhibitor unless approved by the GSK medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2011-03-25 (Actual); Study Completion 2012-03-20 (Actual)

PRIMARY OUTCOMES:
PK data, AEs, changes in laboratory values and vital signs, physical exam, clinical testing and PD data | 21 days

SECONDARY OUTCOMES:
GSK2118436 and its metabolite, PK parameters per protocol following single- and repeat-dose administration of GSK2118436 | 15 days
Change in PD markers including IL-8 in blood, pERK and other markers in tumor biopsies. | 15 days
Correlation between PK, PD, and clinical endpoints. | 15 days
Tumor response as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) | approximately once every 2 months until the end of participation
Urinary ratio of 6-beta-hydroxycortisol to cortisol ratio | 15 days
GSK2118436 PK parameters per protocol with and without food | 15 days
Metabolic profiling in plasma and urine | 15 days
Midazolam PK parameters per protocol | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- Australia (4):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Nedlands, Western Australia

REFERENCES:
- [Background] Hong DS, Vence L, Falchook G, Radvanyi LG, Liu C, Goodman V, Legos JJ, Blackman S, Scarmadio A, Kurzrock R, Lizee G, Hwu P. BRAF(V600) inhibitor GSK2118436 targeted inhibition of mutant BRAF in cancer patients does not impair overall immune competency. Clin Cancer Res. 2012 Apr 15;18(8):2326-35. doi: 10.1158/1078-0432.CCR-11-2515. Epub 2012 Feb 21. PMID 22355009
- [Background] Falchook GS, Long GV, Kurzrock R, Kim KB, Arkenau TH, Brown MP, Hamid O, Infante JR, Millward M, Pavlick AC, O'Day SJ, Blackman SC, Curtis CM, Lebowitz P, Ma B, Ouellet D, Kefford RF. Dabrafenib in patients with melanoma, untreated brain metastases, and other solid tumours: a phase 1 dose-escalation trial. Lancet. 2012 May 19;379(9829):1893-901. doi: 10.1016/S0140-6736(12)60398-5. PMID 22608338
- [Background] Nathanson KL, Martin AM, Wubbenhorst B, Greshock J, Letrero R, D'Andrea K, O'Day S, Infante JR, Falchook GS, Arkenau HT, Millward M, Brown MP, Pavlick A, Davies MA, Ma B, Gagnon R, Curtis M, Lebowitz PF, Kefford R, Long GV. Tumor genetic analyses of patients with metastatic melanoma treated with the BRAF inhibitor dabrafenib (GSK2118436). Clin Cancer Res. 2013 Sep 1;19(17):4868-78. doi: 10.1158/1078-0432.CCR-13-0827. Epub 2013 Jul 5. PMID 23833299
- [Derived] Ouellet D, Gibiansky E, Leonowens C, O'Hagan A, Haney P, Switzky J, Goodman VL. Population pharmacokinetics of dabrafenib, a BRAF inhibitor: effect of dose, time, covariates, and relationship with its metabolites. J Clin Pharmacol. 2014 Jun;54(6):696-706. doi: 10.1002/jcph.263. Epub 2014 Jan 17. PMID 24408395
- [Derived] Carlino MS, Gowrishankar K, Saunders CA, Pupo GM, Snoyman S, Zhang XD, Saw R, Becker TM, Kefford RF, Long GV, Rizos H. Antiproliferative effects of continued mitogen-activated protein kinase pathway inhibition following acquired resistance to BRAF and/or MEK inhibition in melanoma. Mol Cancer Ther. 2013 Jul;12(7):1332-42. doi: 10.1158/1535-7163.MCT-13-0011. Epub 2013 May 3. PMID 23645591
- See also: Results for study 112680 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112680?search=study&study_ids=112680#rs